CLINICAL TRIAL: NCT07224113
Title: Assessment and Educational Intervention to Reduce Ultra-processed Food Consumption in Pediatric Patients With IBD
Status: Recruiting | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Giselle Davila Bernardy, MD, Connecticut Children's Medical Center
Other Study IDs: 25-114
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: IBD; Crohn Disease (CD); Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD); Ultra Processed Food; Nutrition Assessment; DGBI
Keywords: IBD; Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis; Ultra processed food
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD Handout-Only Group: Children and teens with inflammatory bowel disease (Crohn's disease or ulcerative colitis) who receive written nutrition handouts explaining what ultra-processed foods (UPFs) are, common examples, and ways to choose less-processed alternatives.
  Interventions: Behavioral: Handout-Only Intervention
- IBD Handout + Video Group: Children and teens with inflammatory bowel disease who receive both written handouts and a short educational video reinforcing key messages about UPFs, healthy eating, and simple strategies to improve diet quality.
  Interventions: Behavioral: Handout + Video Intervention
- DGBI Control Group: Children and teens with disorders of gut-brain interaction (such as functional abdominal pain or irritable bowel syndrome) who complete the same dietary assessments but do not receive educational materials. This group provides comparison data for baseline dietary patterns.

INTERVENTIONS:
Behavioral: Handout-Only Intervention — Participants receive written nutrition handouts explaining what ultra-processed foods (UPFs) are, how to identify them, and practical strategies to reduce UPF intake.
  Groups: IBD Handout-Only Group
Behavioral: Handout + Video Intervention — Participants receive the same nutrition handouts plus a short educational video reinforcing key messages about UPFs and healthy eating choices.
  Groups: IBD Handout + Video Group

SUMMARY:
This study explores whether simple nutrition education can help children and teens with inflammatory bowel disease (IBD) eat fewer ultra-processed foods (UPFs). UPFs include packaged snacks, sugary drinks, and fast food-items that are high in added sugars, fats, and artificial ingredients. Participants will complete online food recalls to measure what they eat and will then receive either nutrition handouts alone or handouts plus a short educational video about UPFs. Researchers will compare changes in UPF intake between the two groups after several weeks and ask families how useful and acceptable they found the materials. The goal is to identify an effective, practical way to support healthier eating habits and long-term gut health in pediatric IBD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD (Crohn's disease, Ulcerative Colitis, IBD-U) for at least 3 months
* Age 10 through < 22 years at the time of enrollment (i.e., up to the day before the 22nd birthday)
* Followed by a gastroenterologist at Connecticut Children's
* IBD in clinical remission based on calculated PUCAI score <10 or PCDAI score of <10
* Receiving medical infusions at CCMC Infusion Center as part of IBD treatment
* Participants must be on full oral intake and not have major dietary restrictions or require oral nutrition supplements

Exclusion Criteria:

* Following a medically prescribed or restrictive diet such as Crohn's Disease Exclusion Diet (CDED), ketogenic diet, Specific Carbohydrate Diet (SCD), low FODMAP diet, gluten-free diet, paleo, or Whole30.
* Receiving any nutrition through feeding tubes (including nasogastric [NG], nasojejunal [NJ], gastrostomy [G], or gastrojejunostomy [GJ] tubes)
* History of bowel surgery within 3 months of study start affecting ability to sustain normal enteral intake
* Non-English-speaking participants (as translation and short-form consent processes will not be used for this study)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults (ages 8-21 years) with inflammatory bowel disease or a disorder of gut-brain interaction receiving care at Connecticut Children's. Participants will complete dietary recalls and brief surveys to evaluate nutrition education about ultra-processed foods.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Ultra-Processed Food (UPF) Intake | Baseline and follow-up within a 4-12 week window after intervention
  Description: Percent of total daily energy from NOVA Group 4 foods, comparing baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Davila-Bernardy, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No